CLINICAL TRIAL: NCT01313429
Title: Adjuvant Allogeneic Tumor Cell Vaccine With Metronomic Oral Cyclophosphamide and Celecoxib in Patients Undergoing Resection of Sarcomas, Melanomas, Germ Cell Tumors, or Epithelial Malignancies Metastatic to Lungs, Pleura, or Mediastinum
Brief Title: Tumor Cell Vaccine for Patients Undergoing Surgery for Sarcomas, Melanomas, Germ Cell Tumors, or Malignancies That Have Metastasized to the Lungs, Pleura, or Mediastinum
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Per stopping rule if 12 patients underwent immune response analysis after 6 vaccinations and none developed a response, the protocol would stop accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110111; 11-C-0111
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Sarcoma; Melanoma; Epithelial Malignancies; Pleural Malignancies
Keywords: Metastatic Cancer; Cancer Vaccine; Immunotherapy; Adjuvant Therapy; Chest Metastases; Cancer; Melanoma; Lung Cancer; Sarcoma
MeSH Terms: conditions — Sarcoma; Melanoma; Neoplasm Metastasis; Neoplasms; Lung Neoplasms | interventions — Cyclophosphamide; Celecoxib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): tumor cell vaccine administered with chemotherapy
  Interventions: Drug: Cyclophosphamide; Biological: Allogenic tumor Cell Vaccine (K562); Drug: Celecoxib

INTERVENTIONS:
Drug: Cyclophosphamide — 50 mg PO BID for 7 days prior to the first dose of vaccine and then on days 8 through 14, and 22 through 28 of each treatment cycle.
Biological: Allogenic tumor Cell Vaccine (K562) — 4 vaccines consisting of approximately 2.5E7 cells each will be delivered IM every 4 weeks for 6 months. If immune response is detected after first 6 vaccinations, 2 more may be given at 3 month intervals.
Drug: Celecoxib — 400 mg PO BID for 7 days prior to the first dose of vaccine and then on days 1 through 28 of each vaccine cycle.

SUMMARY:
Background:

- Certain types of cancers, including sarcoma and melanoma, have specific antigens (protein molecules) on their surfaces. Research has shown that producing an immune reaction to these antigens may be able to keep tumors from growing by encouraging the immune system to destroy the tumor cells. By creating a vaccine that contains antigens similar to those found on the cancer cells, researchers hope to cause an immune reaction that targets the cancer cells. However, more research is needed to determine the safety and effectiveness of this type of vaccine treatment.

Objectives:

- To determine whether a tumor cell vaccine, given to individuals who have had surgery to remove malignant tumors from the chest, can cause an immune reaction that will prevent the tumors from coming back.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with cancer that has spread to the lungs, pleura, or mediastinum, and have recently had surgery to remove tumors in the chest.

Design:

* Participants will be screened with a physical examination and medical history, as well as blood tests and imaging studies.
* Participants will have the option to have leukapheresis to collect white blood cells for studies on how the body is responding to the vaccine. Participants who agree to have this procedure will have it before the start of treatment and after the sixth and eighth vaccines.
* Seven days before the first vaccine, participants will receive the chemotherapy drugs celecoxib and cyclophosphamide to take twice a day at home.
* Participants will receive the experimental vaccine as an injection in the thigh or arm, and may receive it in two shots depending on how many cells are in each vaccine. Participants will receive a diary to monitor medication doses and side effects, as well as additional cyclophosphamide and celecoxib to take at home as directed by the study.
* Participants will have one vaccine every month for 6 months, and will have regular blood tests and imaging studies. After the sixth vaccine, participants who have successfully responded to the treatment will have two additional vaccines given 3 months apart.
* After the eighth vaccine, participants will have followup visits every 3 months for 1 year and then every 6 months for up to 4 years....

DETAILED DESCRIPTION:
Background:

During recent years, the cancer-testis (CT) antigens (CTA) have emerged as attractive targets for cancer immunotherapy. Whereas malignancies of diverse histologies express a variety of CTAs, immune responses to these antigens appear uncommon in cancer patients, possibly due to low-level, heterogeneous antigen expression, as well as immunosuppressive regulatory T cells. Conceivably, vaccination of cancer patients with allogeneic tumor cells expressing high levels of multiple CTAs in combination with depletion of T regulatory cells will induce broad immunity to these antigens. In order to examine this issue, patients with sarcomas, melanomas, germ cell tumors, or epithelial malignancies metastatic to lungs, pleura or mediastinum will be vaccinated with irradiated K562 erythroleukemia cells expressing GM-CSF (K562-GM) following thoracic metastasectomy. Vaccines will be administered in conjunction with metronomic oral cyclophosphamide (50 mg PO BID x 7d q 14d), and celecoxib (400 mg PO BID). Serologic responses to a variety of recombinant CTAs will be assessed before and after vaccination.

Primary Objectives:

-To assess the safety of K562-GM allogeneic tumor cell vaccines in combination with oral metronomic cyclophosphamide and celecoxib in patients undergoing thoracic metastasectomy.

Eligibility:

* Patients with histologically or cytologically proven sarcoma, melanoma, or epithelial malignancies metastatic to lungs, pleura or mediastinum who can be rendered no clinical evidence of active disease (NED).
* Patients must be 18 years or older with an ECOG performance status of 0 2, without evidence of unstable or decompensated myocardial disease. Patients must have adequate pulmonary reserve evidenced by FEV1 and DLCO equal to or greater than 30% predicted; pCO2 less than 50 mm Hg and pO2 greater than 60 mm Hg on room air ABG; and be on no immunosuppressive medications except inhaled corticosteroids at the time vaccination commences.
* Patients must have a platelet count greater than 100,000, an ANC equal to or greater than 1500 without transfusion or cytokine support, a normal PT, and adequate hepatic function as evidenced by a total bilirubin of <1.5 times upper limits of normal. Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m(2) at the time vaccination commences.

Design:

* Following recovery from thoracic metastasectomy, patients with NED or MRD will be vaccinated via deep subcutaneous injection with 1x10(8) irradiated K562 GM-tumor cells periodically over 6 months.
* Vaccines will be administered in conjunction with metronomic oral cyclophosphamide and celecoxib.
* Systemic toxicities, and immunologic response to therapy will be recorded. Pre and post vaccination serologic responses to a standard panel of CT antigens as well as cell mediated responses to epigenetically-modified autologous EBV-transformed B and autologous tumor cells (if available) will be assessed before and after vaccination.
* Numbers/percentages and function of T regulatory cells in peripheral blood will be assessed before, during, and after vaccinations.
* Patients will be followed in the clinic with routine staging scans until disease recurrence.
* As the exact set of comparisons and analyses to be performed will be determined following completion of the trial, and will be based on limited numbers of patients, the analyses will be considered exploratory and hypothesis generating rather than definitive.
* Approximately 25 patients will be accrued to this trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients with sarcomas, melanomas, germ cell tumors, or epithelial malignancies metastatic to the lungs, mediastinum, or pleura that have no clinical evidence of active disease (NED).
  2. Patients with active disease outside the thorax may be eligible for study once the extrathoracic disease is definitively treated by local modalities such as radiation, surgery, or radiofrequency ablation.
  3. Patients must have received or refused first line standard systemic therapy for their metastases (if applicable).
  4. Patients must be enrolled within 52 weeks following completion of metastasectomy and have shown no evidence of disease during that time.
  5. Patients with intracranial metastases, which have been treated by surgery or radiation therapy may be eligible for study provided there is no evidence of active disease and no requirement for anticonvulsant therapy or steroids following treatment.
  6. Patients must have an ECOG performance status of 0 2.
  7. Patients must be 18 years of age or older due to the unknown effects of immunologic responses to germ cell-restricted gene products during childhood and adolescent development.
  8. Patients must have evidence of adequate bone marrow reserve, hepatic and renal function as evidenced by the following laboratory parameters:

     * Absolute neutrophil count greater than 1500/mm(3)
     * Platelet count greater than 100,000/mm(3)
     * Hemoglobin greater than 8g/dl (patients may receive transfusions to meet this parameter)
     * PT within 2 seconds of the ULN
     * Total bilirubin <1.5 times upper limits of normal
     * Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m(2).
  9. Seronegative for HIV antibody. Note: The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus may be less responsive to the experimental treatment.
  10. Seronegative for active hepatitis B, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
  11. Patients must be aware of the neoplastic nature of their illnesses, the experimental nature of the therapy, alternative treatments, potential benefits, and risks.
  12. Patients must be willing to practice birth control during and for four months following treatment.
  13. Patients must be willing to sign an informed consent.

EXCLUSION CRITERIA:

1. Patients who are initially rendered NED by surgical therapy but exhibit disease progression prior to initiation of vaccination will be excluded from the study.
2. Patients requiring corticosteroids (other than inhaled) will be excluded.
3. Patients with life expectancy less than 12 months will be excluded.
4. Patients receiving warfarin anticoagulation, who cannot be transferred to other agents such as enoxaparin or dabigatran, and for whom anticoagulants cannot be held for up to 24 hours will be excluded.
5. Patients with uncontrolled hypertension (>160/95), unstable coronary disease evidenced by uncontrolled arrhythmias, unstable angina, decompensated CHF (>NYHA Class II), or myocardial infarction within 6 months of study will be excluded.
6. Patients with other cardiac diseases may be excluded at the discretion of the PI following consultation with Cardiology consultants.
7. Patients with any of the following pulmonary function abnormalities will be excluded: FEV, < 30% predicted; DLCO < 30% predicted (postbronchodilator); Oxygen Saturation less than 90% on room air.
8. Pregnant and/or lactating women will be excluded due to the unknown, potentially harmful effects of immune response to CT-X antigens and stem cell proteins that may be expressed in placenta, fetus, and neonates.
9. Patients with active infections, including HIV, will be excluded, due to unknown effects of the vaccine on lymphoid precursors.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-03-04 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Summary of adverse events | 30 days after last vaccine (up to 13 months)
  List of adverse event frequency

SECONDARY OUTCOMES:
Number and description of immunologic responses to a panel of CT antigens in vaccinated patients | After last vaccine
  Number and description of immunologic responses to a panel of CT antigens in vaccinated patients
Paired t test analysis of difference between number and percentage of T reg cells at baseline and at treatment conclusion | After last vaccine
  Assessment of T regs in peripheral blood before and after initiation of CP/celecoxib treatment

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Quiros RM, Scott WJ. Surgical treatment of metastatic disease to the lung. Semin Oncol. 2008 Apr;35(2):134-46. doi: 10.1053/j.seminoncol.2007.12.010. PMID 18396199
- [Background] ALEXANDER J, HAIGHT C. Pulmonary resection for solitary metastatic sarcomas and carcinomas. Surg Gynecol Obstet. 1947 Aug;85(2):129-46. No abstract available. PMID 20253078
- [Background] Pastorino U, Buyse M, Friedel G, Ginsberg RJ, Girard P, Goldstraw P, Johnston M, McCormack P, Pass H, Putnam JB Jr; International Registry of Lung Metastases. Long-term results of lung metastasectomy: prognostic analyses based on 5206 cases. J Thorac Cardiovasc Surg. 1997 Jan;113(1):37-49. doi: 10.1016/s0022-5223(97)70397-0. PMID 9011700
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0111.html